CLINICAL TRIAL: NCT04033497
Title: Treatment Response Assessment Maps (TRAMs) in the Delineation of Radiation Necrosis From Tumor Progression After Stereotactic Radiation in Patients With Brain Metastases: A Prospective Study
Brief Title: Treatment Response Assessment Maps to Delineate Necrosis From Tumor After Stereotactic Radiation in Brain Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Ayal Aizer, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-191
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Brain Tumor
Keywords: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TRAMs I (Experimental): * Magnetic resonance imaging (MRI)-based treatment response assessment maps (TRAMs)
  * Patients with an enlarging lesion in the site of a brain metastasis treated with stereotactic radiation for which neurosurgical resection is planned will undergo preoperative TRAMs
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Magnetic Resonance Imaging will generate imaging of the brain to identify recurrence of tumor.

SUMMARY:
This research study is investigating the value of an imaging study of the brain called an MRI (which stands for magnetic resonance imaging), utilized in unique way, to delineate whether the tumor has recurred or whether radiation changes have occurred after a brain metastasis treated with focused radiation has enlarged.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial.

In this research study, the investigators are utilizing MRIs of the brain with additional post-imaging processing (called Treatment Response Assessment Maps or TRAMs) to try to delineate tumor recurrence from radiation changes. The investigators hope to understand whether such a test may allow future patients to avoid resection entirely.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically or cytologically confirmed solid malignancy of extracranial origin and radiographic evidence of at least one brain metastasis for which stereotactic radiation was utilized in the past. Patients with intracranial pathologic confirmation of a malignancy which originated extracranially but for which extracranial disease has not been biopsied are eligible.
* Participants must have an enlarging lesion in the brain at least 4 months after prior stereotactic radiation to the same site for which neurosurgical resection is planned as routine standard of care.
* Participants must be age 18 years or older.
* Participants must be willing to undergo study procedures.
* The effects of gadolinium / other MRI-based contrast agents on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
* Participants must possess the ability to understand and the willingness to sign a written informed consent document via ink on paper or via an electronic signature medium such as Adobe Sign.

Exclusion Criteria:

* Participants who have a contraindication to MRI (e.g. non compatible implanted metallic device for which MRI is absolutely contraindicated).
* Participants who have chronic kidney disease stage IV-V or end stage renal disease.
* Participants with a history of anaphylactic reactions to gadolinium.
* Pregnant women are excluded from this study because gadolinium-based agents have not been proven to be safe to administer to a developing fetus. Similarly, breastfeeding women will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Within 3 months of study enrollment
  The sensitivity along with 95% exact binomial confidence interval of pre-operative treatment response assessment maps for the identification of viable tumor relative to the gold standard of pathologic review

SECONDARY OUTCOMES:
Specificity | Within 3 months of study enrollment
  The specificity along with 95% exact binomial confidence interval of pre-operative treatment response assessment maps for the identification of viable tumor relative to the gold standard of pathologic review
Positive predictive value | Within 3 months of study enrollment
  The positive predictive value along with 95% exact binomial confidence interval of pre-operative treatment response assessment maps for the identification of viable tumor relative to the gold standard of pathologic review
Negative predictive value | Within 3 months of study enrollment
  The negative predictive value along with 95% exact binomial confidence interval of pre-operative treatment response assessment maps for the identification of viable tumor relative to the gold standard of pathologic review

CONTACTS AND LOCATIONS:
Overall Officials: Ayal Aizer, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu